CLINICAL TRIAL: NCT03200353
Title: Evaluation of Sores Treatment by Oxygenotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NATROX
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Ulcer Venous
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): Each patient included receive the experimental device system NATROX during 3 to 4 weeks
  Interventions: Device: system NATROX (device name)

INTERVENTIONS:
Device: system NATROX (device name) — system NATROX (device name) application on the wounds of lower limbs

SUMMARY:
Patient with chronic wounds are selected to receive NATROX system ; it's a continous diffusion of oxygen therapy delivery system. This one is put on the wound during a consultation at the hospital and will be followed in home medical care. Every 2 days a nurse renew the application at home and patient recharge the system with oxygen every day.

The complete treatment is prescribe for 4 weeks and at the end patient comes to hospital to have a consultation with the doctor.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* accepted to participate
* Patients followed in vascular medicine and entrusted to the home medical care for the bandages of chronic wounds with apathetic ulcers, not presenting of granulation tissue on their surface

Exclusion Criteria:

* infected ulcers
* necrosed ulcers
* Arterial ulcers requiring a revascularisation.
* Ulcers whose surface is superior in 10x10 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
number of patients received the entire treatment (3 to 4 weeks of oxygenotherapy) in home medical care | 4 weeks
  Patients who have received the entire treatment.

SECONDARY OUTCOMES:
percentage of patients who can receive skin graft after the therapy | 1-2 month
  patient eligible to skin graft after the therapy indicate the success of the NATROX system
percentage of patient who stopper the treatment | 4 weeks
  number of patients who have to stop the treatment because of non tolerability among all included patient

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle P LAZARETH, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No